CLINICAL TRIAL: NCT03154463
Title: Analgesic Effect of Three-point Transversus Abdominis Plane Block Compared With Continuous Epidural Infusion for Post-laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Anesthesiology Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes016
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP blocks (Active Comparator): TAP group was received TAP block using ultrasound as a guide and injected on three points on trans abdominal plane using 100 mm stimuplex needle and 0.25% bupivacaine with total volume of 20 ml in each point (with total of 60 ml in three points)
  Interventions: Procedure: TAP Blocks
- continuous epidural infusion (Active Comparator): Epidural group received epidural regional anesthesia in sitting position, with epidural regimen of 0.25% bupivacaine without any adjuvant
  Interventions: Procedure: continuous epidural infusion

INTERVENTIONS:
Procedure: TAP Blocks — TAP blocks were performed using ultrasound as a guide and injected on three points on trans abdominal plane using 100 mm stimuplex needle and 0.25% bupivacaine with total volume of 20 ml in each point (with total of 60 ml in three points)
  Arms: TAP blocks
Procedure: continuous epidural infusion — Continuous epidural infusion was given with epidural regimen of 0.25% bupivacaine without any adjuvant
  Arms: continuous epidural infusion

SUMMARY:
This study aimed to compare the efficacy three-point Transversus Abdominis Plane (TAP) blocks with continuous epidural infusion for alleviating pain post-laparoscopic nephrectomy

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Intravenous (IV) cannula, non-invasive blood pressure monitor, and pulse-oxymetry were set on the subjects in endoscopic room. Vital signs were recorded. Subjects were then randomized into two groups (three-point Transversus Abdominis Plane [TAP] blocks and continuous epidural infusion). The epidural group was received epidural regional anesthesia in sitting position before anesthesia induction, between the first and second lumbar vertebra, with 4 cm depth. The TAP group was received TAP block using ultrasound as a guide and injected in three points on trans abdominal plane using 100 mm stimuplex needle and 0.25% bupivacaine with total volume of 20 ml in each point (with total of 60 ml in three points) after the surgery has ended, before the patient was awake. Subjects were given midazolam 0.05 mg/kg body weight (BW) and fentanyl 1-2 µg/kg BW as premedication. Induction was done using propofol 1-2mg/kg BW. Endotracheal intubation was facilitated using atracurium 0.5 mg/kg BW. General anesthesia was maintained using oxygen, air, and sevoflurane. Mechanical ventilation was set with volume control ventilation, Positive End-Expiratory Pressure (PEEP) 5 cm of water, and oxygen fraction of 30-50%. Respiratory rate was set at certain level until the end-tidal carbon dioxide (CO2) value reached around 35-45 mm Hg. During the surgery, the epidural group only received epidural regimen of 0.25% bupivacaine without any adjuvant, while the TAP group received fentanyl and atracurium if needed. After the surgery ended, subjects were prepared for ventilator weaning and extubation. After the subjects were moved to ward, both groups received additional analgesic consisting of fentanyl with patient-controlled analgesia (PCA) method. Total PCA requirements and visual analog scale (VAS) were recorded in the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were going to donate their kidney with laparoscopic nephrectomy surgery. Patients who undergo surgery with supine position. Patients who agreed to participate in this study.

Exclusion Criteria:

* Subjects with contraindications for TAP blocks or continuous epidural anesthesia, such as infection at the site of injection and blood coagulation disorder

Drop out Criteria:

* Complications such as systemic allergy, anaphylaxis, and cardiac arrest occurs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Total PCA Morphine consumption (in mcg) | Day 1
  Total PCA morphine consumption (in mcg) by subjects at 2,4,6,12, and 24 hours post-operative
Visual Analog Score | Day 1
  Visual analog scale at 2,4,6,12, and 24 hours post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mathuram Thiyagarajan U, Bagul A, Nicholson ML. Pain management in laparoscopic donor nephrectomy: a review. Pain Res Treat. 2012;2012:201852. doi: 10.1155/2012/201852. Epub 2012 Oct 23. PMID 23150820
- [Background] SarinKapoor H, Kaur R, Kaur H. Anaesthesia for renal transplant surgery. Acta Anaesthesiol Scand. 2007 Nov;51(10):1354-67. doi: 10.1111/j.1399-6576.2007.01447.x. PMID 17944639
- [Background] Gulyam Kuruba SM, Mukhtar K, Singh SK. A randomised controlled trial of ultrasound-guided transversus abdominis plane block for renal transplantation. Anaesthesia. 2014 Nov;69(11):1222-6. doi: 10.1111/anae.12704. Epub 2014 Jun 28. PMID 24974901
- [Background] Urigel S, Molter J. Transversus abdominis plane (TAP) blocks. AANA J. 2014 Feb;82(1):73-9. PMID 24654355
- [Background] Bhosale G, Shah V. Combined spinal-epidural anesthesia for renal transplantation. Transplant Proc. 2008 May;40(4):1122-4. doi: 10.1016/j.transproceed.2008.03.027. PMID 18555130
- [Background] Skrekas G, Papalois VE, Mitsis M, Hakim NS. Laparoscopic live donor nephrectomy: a step forward in kidney transplantation? JSLS. 2003 Jul-Sep;7(3):197-206. PMID 14558706
- [Background] Minnee RC, Idu MM. Laparoscopic donor nephrectomy. Neth J Med. 2010 May;68(5):199-206. PMID 20508268
- [Background] Oyen O. Minimally invasive kidney transplantation (MIKT). J Surg Res. 2008 Mar;145(1):4. doi: 10.1016/j.jss.2007.08.001. Epub 2007 Aug 30. No abstract available. PMID 18237747
- [Background] Biglarnia AR, Tufveson G, Lorant T, Lennmyr F, Wadstrom J. Efficacy and safety of continuous local infusion of ropivacaine after retroperitoneoscopic live donor nephrectomy. Am J Transplant. 2011 Jan;11(1):93-100. doi: 10.1111/j.1600-6143.2010.03358.x. PMID 21199350
- [Background] Zhao X, Tong Y, Ren H, Ding XB, Wang X, Zong JY, Jin SQ, Li Q. Transversus abdominis plane block for postoperative analgesia after laparoscopic surgery: a systematic review and meta-analysis. Int J Clin Exp Med. 2014 Sep 15;7(9):2966-75. eCollection 2014. PMID 25356170